CLINICAL TRIAL: NCT05799612
Title: Phase I Study of TH1 Dendritic Cell Immunotherapy for the Treatment of Cutaneous Angiosarcoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cancer Cures 4 Kids (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0018; NCI-2023-02650 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Angiosarcoma
MeSH Terms: conditions — Hemangiosarcoma | interventions — Paclitaxel; RNA, Messenger; peginterferon alfa-2a; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation/Deescalation (Experimental): Participants will receive up to 3 doses of the vaccine (each vaccine is given 2 weeks apart). The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen
  Interventions: Drug: Paclitaxel; Biological: mRNA plus Lysate-loaded Dendritic Cell Vaccine; Drug: PEGYLATED-INTERFERON ALPHA-2A; Drug: Filgrastim

INTERVENTIONS:
Drug: Paclitaxel — Given by IV (vein)
Biological: mRNA plus Lysate-loaded Dendritic Cell Vaccine — Given by IV (vein)
Drug: PEGYLATED-INTERFERON ALPHA-2A — Given by IV (vein)
Drug: Filgrastim — Given by IV (vein)
  Other Names: G-CSF; NeupogenTM

SUMMARY:
To find the highest tolerable dose of an mRNA vaccine that can be safely given to patients with cutaneous angiosarcoma

DETAILED DESCRIPTION:
Objectives:

Primary objective:

•To determine the safety, toxicity, and feasibility of delivering autologous dendritic cells (DCs) loaded with tumor lysate plus mRNA to patients with cutaneous head & neck angiosarcoma as adjuvant therapy.

Secondary objective:

• To assess the recurrence free survival and overall survival in treated patients in order to make initial assessment of activity of this therapeutic approach

Exploratory Objectives:

• To quantitate immune responses in patients who receive autologous DCs loaded with tumor lysate plus mRNA

ELIGIBILITY:
Inclusion criteria:

1. Patients with histologically confirmed cutaneous head & neck angiosarcoma deemed to be potentially resectable and who are deemed to be good candidates for postoperative therapy with radiation and study treatment.
2. Should be willing to undergo biopsy to provide fresh frozen tumor tissue for use in the creation of the vaccine.
3. 18 years of age or older and able to provide informed consent.
4. Adequate kidney, liver, bone marrow function, and immune function, as follows:

   * Hemoglobin ≥ 8.0 gm/dL
   * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
   * Lymphocytes ≥ 500 cells/mm3
   * Platelet count ≥ 75,000 /mm3
   * CD4+ T-cell counts ≥ 200/mm3
   * Glomerular filtration rate (GFR) > 60 mL/min/m2

     * For males = (140 - age[years]) x (body weight [kg]) (72) x (serum creatinine [mg/dL]
     * For females = 0.85 x male value
   * Total bilirubin ≤ 1.5 times upper limit of normal (ULN),
   * Aspartate transaminase AST (SGOT) and alanine aminotransferase ALT (SGPT) ≤ 2.5 times the ULN
   * TSH range between 0.4 - 4.0 mIU / L
   * aPTT or INR ≤ 1.5 × ULN unless subject is receiving anticoagulant therapy. If receiving anticoagulant therapy, patient is eligible as long as prothrombin time, international normalized ratio (INR), or activated partial thromboplastin time is within therapeutic range of intended use of anticoagulants
5. ECOG performance status ≤ 2.

Exclusion criteria:

1. Locally advanced tumors deemed unresectable and/or metastatic tumors
2. Received live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine.
3. Uncontrolled HIV infection with CD4+ <200 c ells/µl or active HBC or HCV disease that requires antiviral therapy.
4. Need for concurrent therapy with corticosteroids or any systemic immunosuppressive agents during the vaccination phase of the study.
5. History of systemic autoimmune disease
6. Female patients who are pregnant, breast feeding, or of childbearing potential without a negative pregnancy test prior to baseline. Male or female patients of childbearing potential unwilling to use contraceptive precautions (refer Table 1) throughout the trial and 3 months following discontinuation of study treatment. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Women of childbearing potential must have a negative serum pregnancy test prior to the first treatment.
7. Concurrent participation on another therapeutic clinical trial.
8. Patients unwilling or unable to comply with the protocol or provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-11-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Ravi, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org